CLINICAL TRIAL: NCT06745921
Title: A Phase 1 Trial to Evaluate the Safety and Immunogenicity of an Inactivated West Nile Virus Vaccine, HydroVax-001B WNV in Healthy Adults
Brief Title: Safety and Immunogenicity of an Inactivated West Nile Virus Vaccine in Healthy Adults
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: 24-0008; 5UM1AI148684-04 (NIH)
Record Dates: First submitted 2024-12-12; First posted 2024-12-20 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-05-13

CONDITIONS: West Nile Viral Infection
Keywords: Healthy Adults; HydroVax-001B WNV; Immunogenicity; Safety; Vaccine; West Nile Virus
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Syringe will be masked
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1A (Experimental): A single, low dose, of 4 mcg of HydroVax-001B West Nile Virus (WNV) vaccine administered intramuscularly once on Day 1, Day 29, and Day 181. N=12
  Interventions: Biological: HydroVax-001B WNV; Other: Sodium Chloride, 0.9%
- Group 1B (Experimental): A single, high dose, of 10 mcg of HydroVax-001B West Nile Virus (WNV)vaccine administered intramuscularly once on Day 1, Day 29, and Day 181. N=12
  Interventions: Biological: HydroVax-001B WNV; Other: Sodium Chloride, 0.9%
- Group 2A (Placebo Comparator): A 0.5 mL dose of placebo, consisting of 0.9 % of NaCl, administered intramuscularly once on Day 1, Day 29, Day 181. N=3
  Interventions: Other: Placebo
- Group 2B (Placebo Comparator): A 0.5 mL dose of placebo, consisting of 0.9 % of NaCl, administered intramuscularly once on Day 1, Day 29, Day 181. N=3
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: HydroVax-001B WNV — A vaccine to West Nile Virus (WNV) that is prepared by propagating naturally attenuated Kunjin strain of WNV on well characterized low-passage Vero cells. The vaccine contains 10 mcg of inactivated purified whole virion WNV formulated in a volume of 0.5 mL/dose with 0.10% aluminum hydroxide, 10% D-sorbitol, 0.001% Polysorbate 80 (Tween80) in 10 mM phosphate-buffer with 350 mM NaCl.
  Arms: Group 1A; Group 1B
Other: Placebo — Placebo
  Arms: Group 2A; Group 2B
Other: Sodium Chloride, 0.9% — 0.9% Sodium Chloride Injection
  Arms: Group 1A; Group 1B

SUMMARY:
A randomized, placebo controlled, double-blind (within dosing group), sequential dose escalation study. This phase 1 trial addresses the urgent need for a vaccine to prevent disease resulting from infection with West Nile virus (WNV), a virus that is primarily spread to people by the bite of an infected mosquito. The purpose of this Phase 1 trial is to evaluate the safety and immunogenicity of the HydroVax-001B WNV vaccine in healthy adult volunteers. The study Population will consist of healthy male and non-pregnant, non-breastfeeding female adults, 18 to 49 years of age, inclusive. Potential participants with a history of prior flavivirus infection or receipt of any flavivirus vaccine or monoclonal antibody, and those who likely had a prior flavivirus infection based on exposure history will be ineligible for the study. Participants will be randomized to receive HydroVax-001B WNV vaccine or placebo in a 12:3 ratio within a dosage group. Participants will be sequentially enrolled into two dosage groups. The primary objective is to assess the safety and reactogenicity of 4 mcg versus 10 mcg dose of the HydroVax-001B WNV vaccine administered intramuscularly (IM) on Days 1, 29 and 181.

DETAILED DESCRIPTION:
A randomized, placebo controlled, double-blind (within dosing group), sequential dose escalation study. This phase 1 trial addresses the urgent need for a vaccine to prevent disease resulting from infection with West Nile virus (WNV), a virus that is primarily spread to people by the bite of an infected mosquito. The purpose of this Phase 1 trial is to evaluate the safety and immunogenicity of the HydroVax-001B WNV vaccine in healthy adult volunteers. The study Population will consist of healthy male and non-pregnant, non-breastfeeding female adults, 18 to 49 years of age, inclusive. Potential participants with a history of prior flavivirus infection or receipt of any flavivirus vaccine or monoclonal antibody, and those who likely had a prior flavivirus infection based on exposure history will be ineligible for the study. Participants will be randomized to receive HydroVax-001B WNV vaccine or placebo in a 12:3 ratio within a dosage group. Participants will be sequentially enrolled into two dosage groups. The primary objective is to assess the safety and reactogenicity of 4 mcg versus 10 mcg dose of the HydroVax-001B WNV vaccine administered intramuscularly (IM) on Days 1, 29 and 181. The secondary objective is to assess immunogenicity of 4 mcg versus 10 mcg dose of HydroVax-001B WNV vaccine given IM on Days 1, 29 and 181 as measured by WNV-specific focus reduction neutralizing test (FRNT50) after each vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Provides written informed consent prior to initiation of any study procedures.
2. Is able to understand and agrees to comply with planned study procedures including being available for all study visits.
3. Agrees to the collection of venous blood per protocol.
4. Is a male or non-pregnant, non-lactating female 18 to 49 years of age, inclusive at time of enrollment.
5. Is in good health.* *Good health is defined by the absence of a medical condition described in the exclusion criteria. If the participant has another current, ongoing medical condition, the condition cannot meet any of the following criteria: (1) was first diagnosed within 3 months of enrollment with a clinically significant condition, in the opinion of investigator that has worsened within 3 months of enrollment; (2) had non-elective surgery, clinically significant medical procedure, or hospitalization within 3 months of enrollment; (3) received new prescription for systemic medication within 30 days of enrollment, unless the new prescription is in the same class of agent or a transition from generic to/from brand name equivalent; or (4) takes medication that may pose a risk to participant's safety or impede assessment of adverse events or study endpoints if they participate in the study.
6. Oral temperature is less than 100.4 degrees Fahrenheit at screening.
7. Pulse is 51 to 100 beats per minute, inclusive at screening.
8. Systolic blood pressure is 90 to 140 mmHg, inclusive at screening.
9. Diastolic blood pressure is 55 to 90 mmHg, inclusive at screening.
10. Screening labs must be within acceptable parameters at screening.*

    *Hematology (white blood cell count [WBC], hemoglobin and platelet count), serum creatinine, blood urea nitrogen, potassium and liver panel (ALT, AST, and total bilirubin) should fall within the normal range of the clinical reference lab. A low creatinine value, low total bilirubin, or a low ALT value are acceptable for trial inclusion as they are not considered to be clinically significant. If screening lab values are within the normal range of the clinical reference lab but fall within the Grade 1 FDA toxicity table range, these will be considered acceptable for enrollment. Urine glucose must be negative and urine protein <1+ (trace urine protein is acceptable) at screening to be eligible for the study. Abnormal urine protein in females on their menses can be repeated after menses is finished.
11. Tests for human immunodeficiency virus (HIV) antigens/antibodies, hepatitis B virus (HBV) surface antigen, and hepatitis C virus (HCV) antibodies must be negative at screening.
12. Females who are of childbearing potential* must agree not to become pregnant during trial.

    *Not of childbearing potential includes post-menopausal females (defined as no menses for at least 12 consecutive months without an alternative medical cause for amenorrhea), or surgically sterile females with documented per volunteer report history of hysterectomy, bilateral oophorectomy, tubal ligation/salpingectomy, or Essure(R) placement and at least 3 months have passed since sterilization procedure.
13. Females of childbearing potential must agree to use an acceptable contraception method* from at least 30 days before the first study vaccination and for the duration of the trial.

    *Acceptable forms of contraception include monogamous relationship with a vasectomized male partner who has been vasectomized for 90 days or more prior to enrollment, use of intrauterine devices, birth control pills, hormonal birth control products that are injectable, implantable (subdermal), transdermal or insertable (vaginal ring), barrier methods with spermicide. Females of childbearing potential who practice abstinence (defined as no heterosexual vaginal-penile intercourse) and agree to practice abstinence consistently for the duration of the study or those who have exclusively non-male sexual relations do not need to use contraception.
14. Females of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test prior to each study vaccination.
15. Has body mass index (BMI) 18.5 kg/m^2 to 34.9 kg/m^2, inclusive.

Exclusion Criteria:

1. Has an acute illness* (with or without fever >/= 38 degrees Celsius [100.4 degrees Fahrenheit]) as determined by the PI or appropriate sub-investigator within 72 hours prior to study product administration.

   *Participants who are afebrile (if applicable) and have either no symptoms or only minor residual symptoms in the 72 hours prior to study product administration can be enrolled if, in the opinion of the site PI or appropriate sub-investigator, the residual symptoms will not interfere with the ability to assess safety parameters as required by the protocol.
2. Has medical disease or condition that, in the opinion of the site PI or appropriate sub-investigator, is a contraindication to study participation.*

   *Including acute, subacute, intermittent, or chronic medical disease or condition that would place the participant an unacceptable risk of injury, render the participant unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the participant's successful completion of this trial.
3. Received systemic anticancer chemotherapy or radiation therapy (cytotoxic) within 3 years prior to enrollment.
4. Has active or recently active (in the 12 months prior to enrollment) neoplastic disease or a history of any hematologic malignancy. Non-melanoma, treated, skin cancers are permitted.
5. Has known allergy to components of the study product.*

   *Including the following: aluminum hydroxide, sorbitol, potassium chloride, sodium chloride and polysorbate80 (Tween80).
6. Has history of idiopathic urticaria.
7. Has history of chronic or acute severe neurologic condition.*

   *Including history of Guillain-Barre syndrome, seizure disorder or epilepsy, Bell's palsy, or disease with any focal neurologic deficits.
8. Has history of alcohol or drug abuse within 5 years prior to study vaccination per investigator's discretion.
9. Has any diagnosis, current or past, of schizophrenia, bipolar disease or other psychiatric diagnosis that may interfere* with participant compliance or safety evaluations.

   *As determined by the site PI or appropriate sub-investigator.
10. Has been hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others within 5 years prior to study vaccination.
11. Has moderate to severe asthma.*

    *Mild, well-controlled asthma may qualify for enrollment as determined by the site PI or appropriate sub-investigator. Cold or exercise induced asthma controlled with inhaled medications other than high - dose inhaled corticosteroids within the past 30 days is permissible. Participants should be excluded if they require daily bronchodilator use or have had an asthma exacerbation requiring oral/parenteral steroid use within the past 30 days or have used theophylline in the past year.
12. Has diabetes mellitus type I or II.*

    *History of gestational diabetes if resolved is acceptable.
13. Is immunosuppressed.*

    *Due to an underlying condition, taking immunomodulatory treatment, or took oral or parenteral (including intra-articular) corticosteroids within the past 30 days or >/= 2 weeks topical corticosteroids of any dose within 30 days prior to study vaccination. Corticosteroid nasal sprays for allergic rhinitis are permissible. Persons using a topical corticosteroid for a limited duration for mild uncomplicated dermatitis such as poison ivy or contact dermatitis may be enrolled the day after their therapy is completed.
14. Have taken high-dose inhaled corticosteroids* within 30 days prior to study vaccination.

    *High-dose defined per reference chart in the National Heart, Lung and Blood Institute Guidelines for the Diagnosis and Management of Asthma (EPR-3).
15. Received or plan to receive a licensed, live vaccine within 30 days before or after each study vaccination.
16. Has received or plans to receive a licensed, inactivated vaccine, including influenza, COVID booster, or allergy desensitization shot, within 14 days before or after study vaccination.
17. Received an experimental agent* within 30 days prior to the study vaccination or expect to receive another experimental agent** during the trial-reporting period.

    *Including vaccine, drug, biologic, device, blood product, or medication.

    **Other than from participation in this trial.
18. Are participating or plan to participate in another clinical trial with an interventional agent* that will be received during the trial-reporting period.

    *Including licensed or unlicensed vaccine, drug, biologic, device, blood product, or medication.
19. Receipt of blood products or immunoglobulin within six months prior enrollment.
20. Donation of a unit of blood within 60 days prior to enrollment or intends to donate blood during the study period.
21. History of WNV infection or other flavivirus infection (e.g., DENV, ZIKV or other flavivirus).
22. History of travel or residency for one month or more in a non-WNV flavivirus-endemic area such as Mexico, Central/South America, the Caribbean, sub-Saharan Africa, South/Southeast Asia, or Polynesia.
23. Plans to visit a flavivirus-endemic country during the study trial period (refer to CDC website for areas with active ZIKV, DENV, YFV, or JEV transmission).
24. History of vaccination with WNV candidate vaccine.
25. History of military service in a flavivirus-endemic region (refer to CDC website for areas with active ZIKV, DENV, YFV, or JEV transmission).
26. History of vaccination against YFV, DENV, TBEV, JEV, ZIKV, WNV, or other licensed or investigational flavivirus vaccines or receipt of monoclonal antibodies against a flavivirus.
27. Attended primary (grade) school in Austria, Germany, Japan, South Korea, India, Thailand, Nepal, Vietnam, or Taiwan (where TBEV vaccine is given).
28. Plan to perform non-routine highly strenuous exercise within 3 days before any clinical safety laboratories.*

    *Safety laboratories are obtained on day of vaccination prior to dosing (i.e. Visit 01, Visit 05, and Visit 11) and Day 15 following each dose of study product (i.e. Visit 04, Visit 08 and Visit 14).
29. Has contraindication to intramuscular vaccination of both upper arms.*

    *Patient with low platelet count or coagulopathy, or someone who is taking oral anticoagulants.
30. Has tattoos, scars, or other marks on both upper arms which would, in the opinion of the investigator, interfere with assessment of the vaccination site.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2025-02-24 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of any unsolicited adverse events (AEs) | Day 1 through Day 29
Frequency of related Grade 3 laboratory toxicities | Day 1 through Day 15
Frequency of related serious adverse events (SAE) overall and in each dose group through the end of the study | Day 1 through study completion, approximately 13 months
  Frequency is the number of discontinuous events
Frequency of solicited local adverse events (AEs) | Day 1 through Day 8
Frequency of solicited systemic adverse events (AEs) | Day 1 through Day 8
Incidence of any unsolicited adverse events (AEs) | Day 1 through Day 29
Incidence of related Grade 3 laboratory toxicities | Day 1 through Day 15
Incidence of related serious adverse events (SAE) overall and in each dose group through the end of the study | Day 1 through study completion, approximately 13 months
  Incidence is the number of participants with an event
Incidence of solicited local adverse events (AEs) | Day 1 through Day 8
Incidence of solicited systemic adverse events (AEs) | Day 1 through Day 8
Severity of any unsolicited adverse events (AEs) | Day 1 through Day 29
Severity of solicited local adverse events (AEs) | Day 1 through Day 8
Severity of solicited systemic adverse events (AEs) | Day 1 through Day 8

SECONDARY OUTCOMES:
Percentage of participants seroconverting | Day 1 through Day 29
  Seroconversion is defined as greater than or equal to 1:10 in FRNT50 titer.
West Nile Virus (WNV)-specific focus reduction neutralizing test (FRNT50) geometric mean titer (GMT) | Day 15 through Day 181

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Louis University Center for Vaccine Development, St Louis, Missouri, United States

DOCUMENTS (1):
  • Informed Consent Form (2024-12-18): https://cdn.clinicaltrials.gov/large-docs/21/NCT06745921/ICF_000.pdf